CLINICAL TRIAL: NCT05594043
Title: A Phase 1, Open-label, Multicenter Study to Assess Safety, Tolerability, PK, and Efficacy of MK-6598 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Tumors
Brief Title: A Study of MK-6598 as Monotherapy and in Combination With Pembrolizumab (MK-3475) in Advanced Solid Tumors (MK-6598-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6598-001; MK-6598-001 (Other: MSD)
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-6598 (Experimental): Participants will receive MK-6598 daily (QD) at escalating dose levels from 50-500 mg for up to a total of 35 cycles (up to approximately 24 months).
  Interventions: Drug: MK-6598
- MK-6598 + Pembrolizumab (Experimental): Participants will receive MK-6598 QD at escalating dose levels from 50-500, plus pembrolizumab 200 mg once every 21-day cycle for up to 35 cycles (up to approximately 24 months).
  Interventions: Drug: MK-6598; Biological: Pembrolizumab

INTERVENTIONS:
Drug: MK-6598 — Oral tablet
Biological: Pembrolizumab — Intravenous (IV) infusion
  Other Names: MK-3475; Keytruda®
  Arms: MK-6598 + Pembrolizumab

SUMMARY:
The purpose of this study is to assess the efficacy and safety and establish a preliminary recommended Phase 2 dose (RP2D) of MK-6598 administered as monotherapy and in combination with pembrolizumab (MK-3475) in adult participants with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically- or cytologically-confirmed advanced/metastatic solid tumor by pathology report and has received, or been intolerant to, all treatment known to confer clinical benefit.
* Has measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the local site investigator/radiology.
* Has one or more discrete malignant lesions that are amenable to a minimum of 2 separate biopsies.
* Has a baseline tumor sample that can be submitted for analysis.
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART).
* A participant assigned male sex at birth who receives MK-6598 must agree to use contraception and should refrain from donating sperm during the specified period(s) of at least 102 days after study interventions.
* A participant assigned female sex at birth is eligible to participate if not pregnant or breastfeeding and at least 1 of the following: not a participant of childbearing potential (POCBP) or a POCBP who agrees to follow the contraceptive guidance during the treatment period and for up to 120 days after study intervention.

Exclusion Criteria:

* Received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention or has not recovered to CTCAE Version 5.0 Grade 1 or better from any AEs that were due to cancer therapeutics administered more than 4 weeks earlier (this includes participants with previous immunomodulatory therapy with residual immune-related AEs).
* Known additional malignancy that is progressing or has required active treatment within 2 years.
* Clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* A severe hypersensitivity (≥Grade 3) reaction to treatment with a monoclonal antibody/components of the study intervention.
* Active infection requiring therapy.
* History of interstitial lung disease.
* History of (noninfectious) pneumonitis that required steroids or current pneumonitis.
* Active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid) is allowed.
* Has known hepatitis B or C infections or known to be positive for hepatitis B surface antigen (HBsAg)/hepatitis B virus (HBV) deoxyribonucleic acid (DNA) or hepatitis C antibody or ribonucleic acid (RNA).
* Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Received prior radiotherapy within 2 weeks of start of study intervention, has radiation-related toxicities requiring corticosteroids, or had a history of radiation pneumonitis.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, CD137), and was discontinued from that treatment due to a ≥Grade 3 immune-related AE (irAE).
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the start of study treatment.
* Has had an allogeneic tissue/solid organ transplant in the last 5 years or has evidence of graft-versus-host disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a Dose-Limiting Toxicity (DLT) Graded Using National Cancer Institute Common Terminology Criteria for Adverse Events (AEs) Version 5.0 | Up to approximately 21 days
  DLT is defined as any of the following toxicities, unless assessed by the investigator to be clearly due to the underlying disease or extraneous causes: Grade (Gr) 4 nonhematologic toxicity (not laboratory); Gr 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia; Gr 4 thrombocytopenia of any duration; Gr 3 thrombocytopenia associated with clinically significant bleeding; Gr 4 anemia regardless of duration; Nonhematologic AE Gr ≥3 in severity, with exceptions; Any Gr 3 or 4 nonhematologic lab abnormality if clinically significant medical intervention is required, or if leads to hospitalization, persists for >72 hours or results in drug-induced liver injury with exceptions; Gr 3 or 4 febrile neutropenia; Prolonged delay (>2 weeks) in initiating Cycle 2 due to treatment-related toxicity; Treatment-related toxicity resulting in study treatment discontinuation during Cycle 1 (C1); Missing >25% of MK-6598 doses as a result of treatment-related AE during C1; Gr 5 toxicity.
Number of Participants Who Experience At Least One AE | Up to approximately 27 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of MK-6598 | Days 1, 8, and 15 of Cycle 1: predose, postdose at 30 minutes (min), 45 min, 60 min, 2 hours (hrs), 6 hrs; Days 2 and 9 of Cycle 1: predose; Day 1 of Cycles 2, 5, 10, 15, 20, 25, 30, and 35: predose
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine AUC.
Minimum Serum Concentration (Cmin) of MK-6598 | Days 1, 8, and 15 of Cycle 1: predose, postdose at 30 min, 45 min, 60 min, 2 hrs, 6 hrs; Days 2 and 9 of Cycle 1: predose; Day 1 of Cycles 2, 5, 10, 15, 20, 25, 30, and 35: predose
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmin
Maximum Serum Concentration (Cmax) of MK-6598 | Days 1, 8, and 15 of Cycle 1: predose, postdose at 30 min, 45 min, 60 min, 2 hrs, 6 hrs; Days 2 and 9 of Cycle 1: predose; Day 1 of Cycles 2, 5, 10, 15, 20, 25, 30, and 35: predose
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmax.
Tumor Phenylpyruvate Concentrations | Days 1, 8, and 15 of Cycle 1: predose, postdose at 30 min, 45 min, 60 min, 2 hrs, 6 hrs; Days 2 and 9 of Cycle 1: predose; Day 1 of Cycles 2, 5, 10, 15, 20, 25, 30, and 35: predose
  Blood samples pre-dose and at multiple timepoints post-dose will be used to determine tumor phenylpyruvate concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- Sanford Cancer Center ( Site 0300), Sioux Falls, South Dakota, United States
- Canada (2):
  - Princess Margaret Cancer Centre ( Site 0101), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal-Unit for Innovative Therapies ( Site 0100), Montreal, Quebec
- Switzerland (3):
  - Hôpitaux Universitaires de Genève (HUG) ( Site 0202), Geneva, Canton of Geneva
  - Ospedale Regionale Bellinzona e Valli ( Site 0200), Bellinzona, Canton Ticino
  - Cantonal Hospital St.Gallen ( Site 0203), Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/